CLINICAL TRIAL: NCT02259673
Title: Mashhad University Medical of Sciences
Brief Title: Effects of Fun Physical Activity on the Interest to Daily Physical Activity and Sarcopenia of Elderly People
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Collaborators: Grudzen, Corita, M.D., MSHS (Individual)
Responsible Party: Principal Investigator, rajabpoor, MUMS, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 920788
Record Dates: First submitted 2014-09-29; First posted 2014-10-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fun exercise (Experimental): effect of fun physical exercise on sarcopenia
  Interventions: Other: Fun exercise
- fun exercise (Experimental): effect of fun physical exercise on interest in exercise
  Interventions: Other: Fun exercise

INTERVENTIONS:
Other: Fun exercise — Intervention group 3 times a week for 20 minutes during 2 months, fun physical exercises (including activities carried out with the use of sports equipment such as beach ball, stretch, bird toys, etc)
Other: fun exercise — Intervention group 3 times a week for 20 minutes during 2 months, fun physical exercises
  (including activities carried out with the use of sports equipment such as beach ball, stretch, bird toys, etc)

SUMMARY:
In this research, the elderly living in nursing homes were selected in two group control and intervention.

Intervention group 3 times a week for 20 minutes during 2 months, fun physical exercises (including activities carried out with the use of sports equipment such as beach ball, stretch, bird toys, etc).

DETAILED DESCRIPTION:
Have of a healthy life with minimal complications in this period. Most important issue in improving the health and quality of life of the elderly is maintain their independence in physical activity. World Health Organization (WHO) is believed that, the first indicator of the health of a society is physical activity of the society.

The studies show that sarcopenia leads to a decrease in the function and increase of disability 2/1 male and 3/1 are older women. sarcopenia leads to some perturbation such as, movement disorders, impaired balance, the incidence of inflammatory disease and dementia. In this reserch, the elderly living in nursing homes were selected in two group control and intervention.

Intervention group 3 times a week for 20 minutes during 2 months, fun physical exercises.

(including activities carried out with the use of sports equipment such as beach ball, stretch, bird toys, etc).

ELIGIBILITY:
Inclusion Criteria:

* age more than 60 year

Exclusion Criteria:

* absence more than 3 session training

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-04 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
interest of daily physical activity | one month
  including activities carried out with the use of sports equipment such as beach ball, stretch, bird toys, etc that will be measured with Exercise Dependence Scale-21 Manual(EDS)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad rajabpoor, Msc student, Study Director — Msc student, Mashhad University Medical of Siences
Locations (1):
- Mashhad University Medical of siences, Mashhad, Iran

REFERENCES:
- [Result] Canga L, Gorelik G, Sterin-Borda L. Diabetes alters the reactivity of myocardium to a thromboxane analogue. Can J Physiol Pharmacol. 1987 Apr;65(4):499-503. doi: 10.1139/y87-085. PMID 2886201
- See also: article cited this sit — http://ncbi.nlm.nih.gov